CLINICAL TRIAL: NCT05193279
Title: A Randomized, Controlled, Dose-finding, Observer-blind, Phase 2/3 Study to Evaluate the Safety, Reactogenicity and Immunogenicity of CpG/Alum-adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccines (SCB-2019 Vaccine) in Children <18 Years of Age
Brief Title: Safety and Immunogenicity of SCB-2019 in Children <18 Years of Age
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was terminated during the EC submission process prior to the enrollment.
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-007
Record Dates: First submitted 2021-12-23; First posted 2022-01-14 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (21):
- SCB-2019/SCB-2019/placebo, 12 to < 18 yrs (Experimental): Day 1 and 22: SCB-2019, Day 43: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Placebo/SCB-2019/SCB-2019, 12 to < 18 years (Experimental): Day 1: placebo, Day 22 and 43: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/placebo/SCB-2019, 12 to < 18 years (Experimental): Day 1 and 43: SCB-2019, Day 22: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Low dose SCB-2019, 5 to < 12 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- Mid dose SCB-2019, 5 to < 12 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- High dose SCB-2019, 5 to < 12 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/SCB-2019/placebo, 5 to < 12 yrs (Experimental): Day 1 and 22: SCB-2019, Day 43: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Placebo/SCB-2019/SCB-2019, 5 to < 12 years (Experimental): Day 1: placebo, Day 22 and 43: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/placebo/SCB-2019, 5 to < 12 years (Experimental): Day 1 and 43: SCB-2019, Day 22: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Low dose SCB-2019, 2 to < 5 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- Mid dose SCB-2019, 2 to < 5 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- High dose SCB-2019, 2 to < 5 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/SCB-2019/placebo, 2 to < 5 yrs (Experimental): Day 1 and 22: SCB-2019, Day 43: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Placebo/SCB-2019/SCB-2019, 2 to < 5 years (Experimental): Day 1: placebo, Day 22 and 43: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/placebo/SCB-2019, 2 to < 5 years (Experimental): Day 1 and 43: SCB-2019, Day 22: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Low dose SCB-2019, birth to < 2 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- Mid dose SCB-2019, birth to < 2 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- High dose SCB-2019, birth to < 2 years (Experimental): Day 1 and 22: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/SCB-2019/placebo, birth to < 2 yrs (Experimental): Day 1 and 22: SCB-2019, Day 43: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019
- Placebo/SCB-2019/SCB-2019, birth to < 2 years (Experimental): Day 1: placebo, Day 22 and 43: SCB-2019
  Interventions: Biological: Candidate vaccine, SCB-2019
- SCB-2019/placebo/SCB-2019, birth to < 2 years (Experimental): Day 1 and 43: SCB-2019, Day 22: placebo
  Interventions: Biological: Candidate vaccine, SCB-2019

INTERVENTIONS:
Biological: Candidate vaccine, SCB-2019 — a recombinant SARS-CoV-2 trimeric S-protein subunit vaccine for COVID-19

SUMMARY:
This is a phase 2/3, randomized, controlled study to assess the reactogenicity, safety and immunogenicity of adjuvanted recombinant SARS-CoV-2 trimeric S-protein subunit vaccine (SCB-2019), when administered as 2-dose vaccination series in children below 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female <18 years of age. Participants will be stratified into different age cohorts (≥12 to < 18 years, ≥5 to < 12 years, ≥2 to < 5 years, and < 2 years of age) based on the age on the day of inclusion.
* Individuals and their legally authorized representative (LAR) are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests and other study procedures.
* Individuals are willing and able to give an assent (if applicable) and their LARs are willing and able to give informed consent on their behalf, prior to screening
* Healthy participants (phase 2 and phase 3) or participants with pre-existing medical conditions who are in a stable medical condition (phase 2)
* For infants (<1-year-old) - born at full term (gestational age ≥37 weeks) and with a normal birth weight (≥2500 grams).
* Female participants of childbearing potential may be enrolled in the study, if the participant has practiced highly effective contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination and has agreed to continue adequate contraception for 3 months after the last vaccination

Exclusion Criteria:

* Individuals with fever >38.0°C [≥ 100.4°F] (irrespective of method used), or any acute illness at baseline (Day 1) or within 3 days prior to randomization.
* Individuals with laboratory-confirmed SARS-CoV-2 infection [as defined by Rapid COVID Antigen Test or an equivalent at Day 1] or with history of laboratory-confirmed/medically-diagnosed COVID-19 (for phase 2 participants only).
* Individuals who have received an investigational or licensed COVID-19 vaccine prior to Day 1, or plan to receive an investigational or licensed COVID-19 vaccine during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease [e.g., malignancy, human immunodeficiency virus (HIV) infection] or immunosuppressive/cytotoxic therapy (e.g., systemic corticosteroids, medications used for cancer chemotherapy, organ transplantation or to treat autoimmune disorders) within 3 months prior to Day 1. Inhaled, intranasal, topical steroids as well as a single dose of systemic steroids, are allowed.
* Individuals with any progressive or severe neurologic disorder, seizure disorder (including febrile seizures) or history of Guillain-Barré syndrome.
* Individuals who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or during the study period.
* Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction
* Individuals who have received any other investigational product within 30 days prior to Day 1 or intend to participate in another clinical study at any time during the conduct of this study.
* Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 28 days after the second (phase 2) or third (phase 3) vaccination.
* Individuals with known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular injection
* Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period
* Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Phase 2, select optimal dose level of SCB-2019 vaccine by age cohort (5-11 years, 2-4 years, and < 2 years), based on safety | 7 days after dose 1 (Day 1-7)
  Proportion of subjects with solicited local and systemic adverse events
Phase 2, select optimal dose level of SCB-2019 vaccine by age cohort (5-11 years, 2-4 years, and < 2 years), based on safety | 7 days after dose 2 (Day 22-28)
  Proportion of subjects with solicited local and systemic adverse events
Phase 2, select optimal dose level of SCB-2019 vaccine in phase 2 by age cohort (5-11 years, 2-4 years, and < 2 years), based on immunogenicity | Day 36
  Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibody (nAb)
Phase 3, non-inferiority (GMT) of SARS-CoV-2 nAb titers of SCB-2019 vaccine when given to participants 5 to < 12 years as compared to young adults (18 to < 25 years) | 21/15 days after second SCB-2019 dose
  GMT of SARS-CoV-2 nAb after 2 doses of SCB-2019 vaccine in participants 5 to 12 years over GMT in participants 18 to < 25 years from CLO-SCB-2019-003 study
Phase 3, non-inferiority (GMT) of SARS-CoV-2 nAb titers of SCB-2019 vaccine when given to participants 2 to < 5 years as compared to young adults (18 to < 25 years) | 21/15 days after second SCB-2019 dose
  GMT of SARS-CoV-2 nAb after 2 doses of SCB-2019 vaccine in participants 2 to 5 years over GMT in participants 18 to < 25 years from CLO-SCB-2019-003 study
Phase 3, non-inferiority (GMT) of SARS-CoV-2 nAb titers of SCB-2019 vaccine when given to participants birth to < 2 years as compared to young adults (18 to < 25 years) | 21/15 days after second SCB-2019 dose
  GMT of SARS-CoV-2 nAb after 2 doses of SCB-2019 vaccine in participants birth to 2 years over GMT in participants 18 to < 25 years from CLO-SCB-2019-003 study

SECONDARY OUTCOMES:
Phase 3, non-inferiority (SCR difference) of SARS-CoV-2 nAb titers of SCB-2019 vaccine when given to participants 5 to < 12 years as compared to young adults (18 to < 25 years) | 21/15 days after second SCB-2019 dose
  Proportion of participants achieving seroconversion for SARS-CoV-2 nAb after 2 doses of SCB-2019 vaccine in participants 5 to < 12 years minus proportion in participants 18 to < 25 years from CLO-SCB-2019-003 study
Phase 3, non-inferiority (SCR difference) of SARS-CoV-2 nAb titers of SCB-2019 vaccine when given to participants 2 to < 5 years as compared to young adults (18 to < 25 years) | 21/15 days after second SCB-2019 dose
  Proportion of participants achieving seroconversion for SARS-CoV-2 nAb after 2 doses of SCB-2019 vaccine in participants 2 to < 5 years minus proportion in participants 18 to < 25 years from CLO-SCB-2019-003 study
Phase 3, non-inferiority (SCR difference) of SARS-CoV-2 nAb titers of SCB-2019 vaccine when given to participants birth to < 2 years as compared to young adults (18 to < 25 years) | 21/15 days after second SCB-2019 dose
  Proportion of participants achieving seroconversion for SARS-CoV-2 nAb after 2 doses of SCB-2019 vaccine in participants birth to < 2 years minus proportion in participants 18 to < 25 years from CLO-SCB-2019-003 study
In phase 2 and 3, GMT of SARS-CoV-2 nAb | Day 1 , 22 and 36 (phase 2) and Day 1, 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, proportion of participants achieving seroconversion for SARS-CoV-2 nAb | Day 22 and 36 (phase 2) and Day 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, GMFR in SARS-CoV-2 nAb | Day 22 and 36 (phase 2) and Day 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, proportion of participants with SARS-CoV-2 nAb above a certain threshold | Day 1 , 22 and 36 (phase 2) and Day 1, 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, GMT of SCB-2019 Binding Antibody | Day 1 , 22 and 36 (phase 2) and Day 1, 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, proportion of participants achieving seroconversion for SCB-2019 binding antibody | Day 22 and 36 (phase 2) and Day 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, GMFR of SCB-2019 binding antibody | Day 22 and 36 (phase 2) and Day 43, 64, 226 and 410 (phase 3)
In phase 2 and 3, proportion of participants with SCB-2019 binding antibody above a certain threshold | Day 1 , 22 and 36 (phase 2) and Day 1, 43, 64, 226 and 410 (phase 3)
In phase 3, reactogenicity of the vaccine as indicated by the occurrence of solicited local and systemic reactions | 7 days after dose 1 (Day 1-7), dose 2 (Day 22-Day 28) and Dose 3 (Day 43-49)
  In phase 3, proportion of participants with local and systemic AEs
Phase 2 and 3, safety of the vaccine in terms of occurrence of unsolicited adverse events | Up to 21 days after the last vaccination
  Proportion of subjects with unsolicited adverse events
Phase 2 and 3, safety of the vaccine in terms of occurrence of MAAEs, SAEs, adverse events leading to discontinuation from study, and AESIs. | During the entire study period
  Proportion of participants with any adverse events in this category.

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Clínica de la Costa Ltda, Barranquilla
  - Centro de Estudios en Infectología Pediátrica S.A.S. - CEIP S.A.S., Cali